CLINICAL TRIAL: NCT05369117
Title: To Evaluate Whether the Clinical Efficacy of Laparoscopic Lymph Node Dissection With Indocyanine Green Tracer is Better Than Without Indocyanine Green Tracer
Brief Title: Application of Indocyanine Green Labeled Fluorescent Laparoscopy in Proximal Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangyong Zhang (Other)
Responsible Party: Sponsor-Investigator, Guangyong Zhang, Director of General Surgery department, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(021)
Record Dates: First submitted 2022-04-25; First posted 2022-05-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer
Keywords: Indocyanine green
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indocyanine green labeled fluorescent laparoscopy (Experimental): The experimental group was marked with indocyanine green, while the control group was not marked with indocyanine green
  Interventions: Behavioral: indocyanine green labeled fluorescent laparoscopy
- The pathological staging (Experimental): They were grouped by different pathological stages
  Interventions: Behavioral: indocyanine green labeled fluorescent laparoscopy

INTERVENTIONS:
Behavioral: indocyanine green labeled fluorescent laparoscopy — indocyanine green fluorescence labeling was performed under gastroscope before surgery and internal jugular vein puncture was performed routinely for better fluid replenishment after surgery

SUMMARY:
Recently, laparoscopic gastrectomy has been gradually accepted by surgeons worldwide for gastric cancer treatment. Complete dissection of the lymph nodes and the establishment of the surgical margin are the most important considerations for curative gastric cancer surgery. Previous studies have demonstrated that indocyanine green (ICG)-traced laparoscopic gastrectomy significantly improves the completeness of lymph node dissection. However, it remains difficult to identify the tumor location intraoperatively for gastric cancers that are staged ≤T3. Here, the investigatorsinvestigated the feasibility of ICG fluorescence for lymph node mapping and tumor localization during totally laparoscopic distal gastrectomy.Preoperative and perioperative data from consecutive patients with gastric cancer who underwent a laparoscopic proximal gastrectomy were collected and analyzed. The investigators want to know if near-infrared fluorescence imaging with ICG can be successfully used in laparoscopic proximal gastrectomy, and if it contributes to both the completeness of D2 lymph node dissection and confirmation of the gastric transection line. The application of ICG labeled near infrared imaging fluorescence laparoscopic technology is still in the stage of exploration and experience accumulation, and it needs to be comprehensively evaluated through a large number of prospective randomized controlled studies.

DETAILED DESCRIPTION:
Recently, laparoscopic gastrectomy has been gradually accepted by surgeons worldwide for gastric cancer treatment. Complete dissection of the lymph nodes and the establishment of the surgical margin are the most important considerations for curative gastric cancer surgery. Previous studies have demonstrated that indocyanine green (ICG)-traced laparoscopic gastrectomy significantly improves the completeness of lymph node dissection. However, it remains difficult to identify the tumor location intraoperatively for gastric cancers that are staged ≤T3. Here, the investigatorsinvestigated the feasibility of ICG fluorescence for lymph node mapping and tumor localization during totally laparoscopic distal gastrectomy.Preoperative and perioperative data from consecutive patients with gastric cancer who underwent a laparoscopic proximal gastrectomy were collected and analyzed. The investigators want to know if near-infrared fluorescence imaging with ICG can be successfully used in laparoscopic proximal gastrectomy, and if it contributes to both the completeness of D2 lymph node dissection and confirmation of the gastric transection line. The application of ICG labeled near infrared imaging fluorescence laparoscopic technology is still in the stage of exploration and experience accumulation, and it needs to be comprehensively evaluated through a large number of prospective randomized controlled studies.By recruiting patients and signing informed consent, randomized control was used to divide patients into the experimental group (fluorescently labeled fluorescently laparoscopic proximal gastric cancer surgery) and the control group (fluorescently labeled fluorescently laparoscopic proximal gastric cancer surgery). In the experimental group, indocyanine green fluorescence labeling was performed under gastroscope before surgery and internal jugular vein puncture was performed routinely for better fluid replenishment after surgery. Lymph nodes and diseased stomach tissues were collected during operation. Postoperative assessment was made for ICU support, routine acid-suppressing therapy, prophylactic antibiotics, analgesia, and nausea suppression. The patients were followed up for 3 years. The primary outcome was 3-year disease-free survival, and the secondary outcome was lymph node positive rate, early complication rate and surgical mortality. The investigators plan to obtain more precise evidence-based medical evidence through this project.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old < age < 75 years old
2. The primary gastric lesion was pathologically diagnosed as proximal gastric adenocarcinoma by endoscopic biopsy (papillary adenocarcinoma PAP, tubular adenocarcinoma TUB, mucinous adenocarcinoma MUC, signed-ring cell carcinoma SIG, poorly differentiated adenocarcinoma POR)
3. Preoperative clinical staging was CT1-4A, N-/+, and M0, according to AJCC-8th TNM tumor staging
4. No distant metastasis was found in preoperative examination, and the tumor did not directly invade pancreas, spleen or other adjacent organs
5. ECOG physical status score 0/1 before surgery Preoperative ASA score I-III

(7) Informed consent of patients

Exclusion Criteria:

1. Suffering from severe mental illness
2. Severe complications cannot tolerate surgery
3. Simultaneous surgical treatment of other diseases is required
4. History of gastric surgery (including ESD/EMR for gastric cancer)
5. Tumors involving esophagus or duodenum were confirmed preoperatively
6. Neoadjuvant therapy has been implemented
7. Leather stomach
8. Refusing laparoscopic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Three-year disease-free survival rate | Through study completion，an average of 3 years
  To evaluate the difference of 3-year disease-free survival rate between the experimental group and the control group

SECONDARY OUTCOMES:
lymph node positive rate | up to 1 week
  To evaluate the difference oflymph node positive rate between the experimental group and the control group
Incidence of early complications | up to 1 week
  The incidence of lymphatic leakage, shock and gastric stump leakage were used as secondary outcome measures
operative mortality | up to 24 hours
  To investigate whether the mortality of laparoscopic proximal gastric cancer surgery marked with indocyanine green was lower than that of the control group

IPD SHARING:
Plan to Share IPD: No